CLINICAL TRIAL: NCT01164618
Title: The Biology of Chronic Preconditioning: Genomic and Physiologic Mechanisms of Response
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Andrew Redington, Head, Heart Centre-Cardiology Division, The Hospital for Sick Children
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1000015862
Record Dates: First submitted 2010-07-14; First posted 2010-07-16 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-08

CONDITIONS: Ischemic Preconditioning
Keywords: pediatrics; Remote ischemic preconditioning
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): The subjects in this arm will begin on the daily remote ischemic preconditioning (RIPC) protocol for 10 days. After a 21 day washout period they will then crossover to 10 days of daily exercise.
  Interventions: Procedure: Remote ischemic preconditioning (RIPC); Other: Exercise
- Group 2 (Experimental): The subjects in this arm will begin on the exercise protocol for 10 days. After a 21 day washout period they will then crossover to 10 days of daily remote ischemic preconditioning (RIPC).
  Interventions: Procedure: Remote ischemic preconditioning (RIPC); Other: Exercise

INTERVENTIONS:
Procedure: Remote ischemic preconditioning (RIPC) — RIPC will be induced using a standard blood pressure cuff and hand anaeroid sphygmomanometer, on the right arm. The subject will be seated, the blood pressure cuff placed on the arm and inflated to a pressure of 200mmHg for 5 minutes (ischemia). The cuff will then be deflated for 5 minutes (reperfusion) completing one cycle of ischemia reperfusion. A total of 4 inflation and deflation cycles will be applied. This protocol of RIPC will be applied daily, for 10 consecutive days.
Other: Exercise — Subjects will then undergo exercise daily, for 10 consecutive days. A chronic high-intensity interval exercise training protocol standardized to subjects' aerobic power (VO¬2max) will be used. Each exercise session will consist of a 5 min warm-up period followed by 4 sets of 2 min high intensity intervals interspersed with 3 min recovery periods.

SUMMARY:
The purpose of this study is to assess the effects of repeated RIPC and exercise, on exercise performance, skeletal muscle responses and circulating cellular and humoral biology in humans

DETAILED DESCRIPTION:
Remote ischemic preconditioning (RIPC) results in a powerful and widespread protective effect against subsequent prolonged ischemia-reperfusion (IR) injury of distant organs and systemic inflammatory responses, both of which are key elements in the evolution of local and multiorgan effects of many clinical IR syndromes. The signal transduction within the target organ to generate ischemia tolerance, and the effects of RIPC on systemic anti-inflammatory pathways, however, remain to be elucidated fully. Particularly, data regarding the mechanisms of 'second window' protection (a resurgence of protection 24-72 hrs after the initial RIPC stimulus) is scant; even less is known of the effects of repeated RIPC, and a potential 'third window' of protection. Our preliminary data and several recent publications have shown that the biology of RIPC and exercise show considerable overlap. This research has raised the possibility of a reciprocal effect between RIPC and exercise, with chronic exercise being a model of the potential effects of 'chronic preconditioning'. This is relevant, as repeated RIPC might be a strategy to improve exercise function in those with limited exercise tolerance e.g. heart failure.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years,
2. Informed consent

Exclusion Criteria:

1. Contraindication to exercise,
2. Vigorous aerobic/anaerobic exercise in duration of ≥15 minutes during the 21 days prior to commencement of the study, or either of the RIPC or exercise protocol arms,
3. Overt viral or bacterial infection in the 10 days prior to commencement of the study, or during either of the RIPC or exercise protocol arms,
4. Alcohol and/or caffeine consumption in the 10 days prior to, or at any time during the study period
5. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2010-05; Primary Completion 2013-02 (Actual); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Ischemia-reperfusion injury tolerance | Day 1 of the Excercise intervention
  This will be done to assess whether chronic preconditioning in humans generates a circulating effector(s) responsible for the generation of cardioprotection in our mouse model of ischemia-reperfusion injury.
  This measure will be compared over time within groups and between groups.
Ischemia-reperfusion injury tolerance | Day 1 of the RIPC intervention
  This will be done to assess whether chronic preconditioning in humans generates a circulating effector(s) responsible for the generation of cardioprotection in our mouse model of ischemia-reperfusion injury.
  This measure will be compared over time within groups and between groups.
Ischemia-reperfusion injury tolerance | Day 2 of the Excercise intervention
  This will be done to assess whether chronic preconditioning in humans generates a circulating effector(s) responsible for the generation of cardioprotection in our mouse model of ischemia-reperfusion injury.
  This measure will be compared over time within groups and between groups.
Ischemia-reperfusion injury tolerance | Day 2 of the RIPC intervention
  This will be done to assess whether chronic preconditioning in humans generates a circulating effector(s) responsible for the generation of cardioprotection in our mouse model of ischemia-reperfusion injury.
  This measure will be compared over time within groups and between groups.
Ischemia-reperfusion injury tolerance | Day 10 of the Excercise intervention
  This will be done to assess whether chronic preconditioning in humans generates a circulating effector(s) responsible for the generation of cardioprotection in our mouse model of ischemia-reperfusion injury.
  This measure will be compared over time within groups and between groups.
Ischemia-reperfusion injury tolerance | Day 10 of the RIPC intervention
  This will be done to assess whether chronic preconditioning in humans generates a circulating effector(s) responsible for the generation of cardioprotection in our mouse model of ischemia-reperfusion injury.
  This measure will be compared over time within groups and between groups.

SECONDARY OUTCOMES:
Change in skeletal muscle metabolic parameters metabolism as measured by 31P-MRS and BOLD fMRI over time within groups and between groups | Days 1, 2 and 10 days of each intervention (RIPC and Excercise)
Neutrophil Function - adhesion, phagocytotic index, and superoxide production over time within groups and between groups | Days 1, 2 and 10 of each intervention (RIPC and Excercise)
Neutrophil Gene Expression over time within groups and between groups | Days 1, 2 and 10 of each intervention (RIPC and Excercise)
Ischemia-reperfusion injury tolerance | Days 1, 2 and 10 of each intervention (RIPC and Excercise)
  We will assess whether chronic preconditioning in humans generates a circulating effector(s) responsible for the generation of cardioprotection in our mouse model of ischemia-reperfusion injury.
Exercise Capacity (VO2max) over time within groups and between groups | Day 10 of each intervention (RIPC and Exercise)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Redington, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada